CLINICAL TRIAL: NCT07106125
Title: Trial of Antibiotic Strategies for Kidney Transplant Recipients
Brief Title: Antibiotics for Kidney Transplant Recipients
Acronym: TASK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25-44366
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Kidney Transplant; Urinary Tract Infection(UTI); Antibiotic Prophylaxis; Remote Patient Monitoring; Feasibility Pilot Study
Keywords: kidney transplant; UTI prevention; antibiotic prophylaxis; decentralized trial; remote clinical trial
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug (Experimental): TMP-SMX
  Interventions: Drug: Trimethoprim-Sulfamethoxazole (TMP-SMX)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole (TMP-SMX) — Kidney transplant recipients will continue to take TMP-SMX daily from months 6-12 after transplant
  Arms: Drug
Other: Usual Care — Participants will take a placebo from months 6-12 after transplant and continue to receive all standard usual care related to their kidney transplant status
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if a common antibiotic called trimethoprim-sulfamethoxazole (TMP-SMX) can help prevent urinary tract infections (UTIs) in children and young adults who recently had a kidney transplant. Most people take TMP-SMX for about 6 months after getting a kidney transplant. In this study, researchers want to see what happens if people keep taking it for 6 more months.

The main questions this study is asking are:

* Does TMP-SMX lower the number of UTIs in the first year after transplant?
* What side effects or problems do participants have while taking TMP-SMX?

Researchers will compare TMP-SMX to a placebo (a look-alike pill that does not contain any medication) to see if TMP-SMX works to prevent UTIs.

Participants will:

* Take either TMP-SMX or a placebo pill by mouth every day for 6 months
* Have three visits to touch base with the study team about any issues
* Complete short monthly online surveys about any symptoms or side effects
* Share blood and urine test results from their regular transplant clinic visits

ELIGIBILITY:
Inclusion Criteria:

* Must be able to take capsules orally
* Kidney transplant performed at a UCSF facility within the last 6 months
* Most recent glomerular filtration rate (GFR) >30 mL/min/1.73 m2
* Tolerated initial 6 months of post-transplant TMP-SMX (defined as no intentional periods of TMP-SMX cessation in first 6 months after transplant due to hyperkalemia, allergic reaction, or unexpected/excessive neutropenia)
* Considered "high risk for UTI" after kidney transplant, as defined by one or more of the following: (1) Congenital anomaly of kidney/urinary tract as kidney failure etiology, (2) Diagnosis of neurogenic bladder and/or use of clean intermittent catheterization and/or nightly continuous urinary drainage, (3) Diabetes mellitus (diagnosed either prior to or new-onset after transplant), (4) History of recurrent UTIs as diagnosed by a provider prior to transplant, (5) Occurrence of any UTI in first 6 months after transplant, (6) Delayed graft function (defined as need for dialysis within 7 days of transplant)

Exclusion Criteria:

* History of intolerance or allergy to trimethoprim (TMP) and/or sulfamethoxazole (SMX)
* History of UTI due to a TMP-SMX-resistant organism in the first 6 months after transplant
* Moderate or severe neutropenia (absolute neutrophil count <1,000 cells/μL) on most recent bloodwork available at the time of recruitment
* Uncontrolled hyperkalemia (serum potassium ≥5.0 mEq/L) on most recent bloodwork available at the time of recruitment
* Provider-determined/documented need for either continuation or discontinuation of TMP-SMX prophylaxis that would preclude the patient's randomization
* Current pregnancy
* Incarcerated individuals/prisoners
* Inability to provide informed consent or assent, and no legally authorized representative available

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Agreement Between Participant Self-Report and Medical Records on Clinical Events (Measured by Cohen's Kappa) | From enrollment to the end of the study drug period (6 months)
  The investigators will look at how closely participants' self-reports of events (urinary tract and associated infections, acute kidney injury events, and hospitalizations) match what is identified through their electronic health records. To do this, the investigators will use a statistical tool called Cohen's kappa, which shows how much agreement there is between the two sources.
Number of Participants Who Enroll After Screening | Baseline/Study Day 1 (i.e., date that informed consent is signed for those who choose to participate)
  The investigators will track how many people decide to join and how many people decline to join the study after completing the screening process.
Medication Adherence Assessed by Self-Report | From enrollment to the end of the study drug period (6 months)
  The investigators will ask participants how often they are taking the pills as directed, through monthly surveys and at all study visits.
Trial Retention | From enrollment to the end of the study drug period (6 months)
  The investigators will keep track of how many participants complete the last study visit

SECONDARY OUTCOMES:
Event Rate of All-Cause Hospitalizations by Treatment Arm | From enrollment through the end of the study period (12 months)
  The investigators will keep track of when participants are hospitalized, using feedback from participants themselves (for the first 6 months) as well as data from their electronic medical records (for 6 additional months, for a total of 12 months). Event rates will be used to compare outcomes between the treatment (TMP-SMX continuation) and placebo arms.
Urinary Tract Infections by Treatment Arm | From enrollment to the end of the study period (12 months)
  The investigators will keep track of when participants report having a urinary tract infection, using feedback from participants themselves (for the first 6 months) as well as data from their electronic medical records (for 6 additional months, for a total of 12 months). Event rates will be used to compare outcomes between the treatment (TMP-SMX continuation) and placebo arms.
Acute Kidney Injury Events by Treatment Arm | From enrollment to the end of the study period (12 months)
  The investigators will keep track of when participants report having acute kidney injury events, using feedback from participants themselves (for the first 6 months) as well as data from their electronic medical records (for 6 additional months, for a total of 12 months). Event rates will be used to compare outcomes between the treatment (TMP-SMX continuation) and placebo arms.
Adverse Events by Treatment Arm | From enrollment to the end of the study drug period (6 months)
  The investigators will keep track of when participants report side effects and adverse events, using feedback from participants themselves as well as data from their electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Bicki, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations, the access, distribution, and reuse of the resulting scientific data will not be permitted. The study involves minors and a sample size that may be prone to "small cells" (using the Centers for Medicare and Medicaid definition of <10 individuals with certain characteristics). We will not share individual-participant level data.